CLINICAL TRIAL: NCT01162031
Title: Phase II Study of Bortezomib (VELCADE) for the Treatment of Relapsed or Refractory T-cell Prolymphocytic Leukemia
Brief Title: Phase II Study of VELCADE for Relapsed or Refractory T-cell Prolymphocytic Leukemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no accrual
Sponsor: Stanford University (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-15361; X05278 (Other: Millennium Pharmaceuticals); SU-09232008-1304 (Other: Stanford University); HEMTPLL0001 (Other: OnCore)
Record Dates: First submitted 2010-07-12; First posted 2010-07-14 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Leukemia; Acute Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Velcade — IV
  Other Names: Bortezomib

SUMMARY:
We hope to learn more about the clinical efficacy of bortezomib in T-cell prolymphocytic leukemia. Patients will be selected as a possible participant in this study because they have a bone marrow disorder known as T-cell prolymphocytic leukemia (T-cell PLL) which does not tend to respond well to conventional treatment with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:Each patient must meet all of the following inclusion criteria to be enrolled in the study:

* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male subject agrees to use an acceptable method for contraception for the duration of the study.
* Bilirubin: <2.0 x Upper limit of normal (ULN)/ Alanine Transaminase (ALT): <3.0 x ULN (<5x ULN if hepatic compromise is present).
* Eastern Cooperative Group (ECOG) 0-2.
* Confirmed diagnosis of T-cell PLL according to the WHO classification.
* Confirmed prior therapy to which the subject was documented to be either refractory or has relapsed since treatment and first documented response.

Exclusion Criteria:Patients meeting any of the following exclusion criteria are not to be enrolled in the study.

* Patient has a platelet count of <30' 10 9/L within 14 days before enrollment.
* Patient has an absolute neutrophil count of <1.0 ´ 10 9/L within 14 days before enrollment.
* Patient has ³Grade 2 peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see section 8.4), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to bortezomib, boron or mannitol.
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum b-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has received other investigational drugs with 14 days before enrollment.
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Patients with uncontrolled intercurrent illness, active or uncontrolled infections, or a fever >38.5c on the day of scheduled dosing.
* Patients with serious illnesses, medical conditions, or other medical history, including laboratory results, which, in the investigator's opinion, would be likely to interfere with a patient's participation in the study, or with the interpretation of the results.
* Any condition (e.g., known or suspected poor compliance, psychological instability, geographical location, etc) that, in the judgment of the investigator, may affect the patient's ability to sign the informed consent and undergo study procedures.
* Any condition that will put the patient at undue risk or discomfort as a result of adherence to study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Assess the clinical activity, as represented by the overall response rate (complete response + partial response), of bortezomib in patients with relapsed or refractory T-cell prolymphocytic leukemia (PLL) | 1 year

SECONDARY OUTCOMES:
prolymphocytic leukemia (PLL) | 1 year
Evaluate time to progression in patients with T-cell prolymphocytic leukemia (PLL) | 1 year
Evaluate the 1-year progression free survival (PFS), and 1-year overall survival (OS) in patients with T-cell prolymphocytic leukemia (PLL) treated with Velcade compared to historical controls | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Carneiro de Medeiros, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States